CLINICAL TRIAL: NCT05050084
Title: Parallel Phase III Randomized Trials of Genomic-Risk Stratified Unfavorable Intermediate Risk Prostate Cancer: De-Intensification and Intensification Clinical Trial Evaluation (GUIDANCE)
Brief Title: Two Studies for Patients With Unfavorable Intermediate Risk Prostate Cancer Testing Less Intense Treatment for Patients With a Low Gene Risk Score and Testing a More Intense Treatment for Patients With a Higher Gene Risk Score, The Guidance Trial
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: NRG Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NRG-GU010; NCI-2021-08760 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); NRG-GU010 (Other: NRG Oncology); NRG-GU010 (Other: CTEP); U10CA180868 (NIH)
Record Dates: First submitted 2021-09-09; First posted 2021-09-20 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Prostate Adenocarcinoma
MeSH Terms: interventions — bicalutamide; Buserelin; darolutamide; acetyl-2-naphthylalanyl-3-chlorophenylalanyl-1-oxohexadecyl-seryl-4-aminophenylalanyl(hydroorotyl)-4-aminophenylalanyl(carbamoyl)-leucyl-ILys-prolyl-alaninamide; Flutamide; Salicylic Acid; Goserelin; histrelin; Leuprolide; Radiotherapy; Radiation; relugolix; Triptorelin Pamoate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Arm I (RT) (Experimental): Patients undergo radiation therapy (RT) using a recognized regimen (2-3 days a week or 5 days a week for 2-11 weeks) in the absence of disease progression or unacceptable toxicity.
  Interventions: Radiation: Radiation Therapy
- Arm II (RT, ADT) (Experimental): Patients undergo RT as Arm I. Patients also receive androgen deprivation therapy (ADT) consisting of leuprolide, goserelin, buserelin, histrelin, triptorelin, degarelix, or relugolix at the discretion of the treating physician, for 6 months in the absence of disease progression or unacceptable toxicity. Patients may also receive bicalutamide or flutamide for 0, 30 or 180 days.
  Interventions: Drug: Bicalutamide; Drug: Buserelin; Drug: Degarelix; Drug: Flutamide; Drug: Goserelin; Drug: Histrelin; Drug: Leuprolide; Radiation: Radiation Therapy; Drug: Relugolix; Drug: Triptorelin
- Arm III (RT, ADT) (Experimental): Patients receive treatment as in Arm II.
  Interventions: Drug: Bicalutamide; Drug: Buserelin; Drug: Degarelix; Drug: Flutamide; Drug: Goserelin; Drug: Histrelin; Drug: Leuprolide; Radiation: Radiation Therapy; Drug: Relugolix; Drug: Triptorelin
- Arm IV (RT, ADT, darolutamide) (Experimental): Patients receive RT and ADT as in Arm II. Patients also receive darolutamide PO BID on days 1-90. Treatment repeats every 90 days for up to 2 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Buserelin; Drug: Darolutamide; Drug: Degarelix; Drug: Goserelin; Drug: Histrelin; Drug: Leuprolide; Radiation: Radiation Therapy; Drug: Relugolix; Drug: Triptorelin

INTERVENTIONS:
Drug: Bicalutamide — Drug
  Other Names: Casodex; Cassotide; Cosudex; ICI 176,334; ICI 176334; Utamide
  Arms: Arm II (RT, ADT); Arm III (RT, ADT)
Drug: Buserelin — Drug
  Other Names: 6-[O-(1,1-Dimethylethyl)-D-serine]-9-(N-ethyl-L-prolinamide)-10-deglycinamide-luteinizing Hormone-releasing Factor (Pig); BSRL; Busereline; Etilamide; HOE 766; HOE-766; HOE766; ICI 123215; ICI-123215; ICI123215; S74 6766; S74-6766; S746766; Tiloryth
  Arms: Arm II (RT, ADT); Arm III (RT, ADT); Arm IV (RT, ADT, darolutamide)
Drug: Darolutamide — Given PO
  Other Names: Antiandrogen ODM-201; BAY 1841788; BAY-1841788; BAY1841788; Nubeqa; ODM 201; ODM-201; ODM201
  Arms: Arm IV (RT, ADT, darolutamide)
Drug: Degarelix — Drug
  Other Names: ASP 3550; ASP-3550; ASP3550; FE 200486; FE-200486; FE200486; Firmagon
  Arms: Arm II (RT, ADT); Arm III (RT, ADT); Arm IV (RT, ADT, darolutamide)
Drug: Flutamide — Drug
  Other Names: 4'-Nitro-3'-trifluoromethylisobutyranilide; Apimid; Cebatrol; Chimax; Cytomid; Drogenil; Euflex; Eulexine; Flucinom; Flucinome; Flugerel; Fluken; Flulem; FLUT; Fluta-Gry; Flutabene; Flutacan; Flutamex; Flutamin; Flutan; Flutaplex; Fugerel; Grisetin; Niftolide; Oncosal; Profamid; Propanamide, 2-Methyl-N-(4-nitro-3-(trifluoromethyl)phenyl)-; Prostacur; Prostadirex; Prostica; Prostogenat; Sch 13521; Tafenil; Tecnoflut; Testotard
  Arms: Arm II (RT, ADT); Arm III (RT, ADT)
Drug: Goserelin — Drug
  Other Names: ICI-118630
  Arms: Arm II (RT, ADT); Arm III (RT, ADT); Arm IV (RT, ADT, darolutamide)
Drug: Histrelin — Drug
  Arms: Arm II (RT, ADT); Arm III (RT, ADT); Arm IV (RT, ADT, darolutamide)
Drug: Leuprolide — Drug
  Other Names: Leuprorelin
  Arms: Arm II (RT, ADT); Arm III (RT, ADT); Arm IV (RT, ADT, darolutamide)
Radiation: Radiation Therapy — Undergo RT
  Other Names: Cancer Radiotherapy; Energy Type; ENERGY_TYPE; Irradiate; Irradiated; Irradiation; Radiation; Radiation Therapy, NOS; Radiotherapeutics; Radiotherapy; RT; Therapy, Radiation
Drug: Relugolix — Drug
  Other Names: N-(4-(1-((2,6-Difluorophenyl)methyl)-5-((dimethylamino)methyl)-1,2,3,4-tetrahydro-3-(6-methoxy-3-pyridazinyl)-2,4-dioxothieno(2,3-d)pyrimidin-6-yl)phenyl)-N'-methoxyurea; Orgovyx; Relumina; TAK 385; TAK-385; TAK385
  Arms: Arm II (RT, ADT); Arm III (RT, ADT); Arm IV (RT, ADT, darolutamide)
Drug: Triptorelin — Drug
  Other Names: 6-D-Tryptophan-LH-RH; 6-D-Tryptophanluteinizing Hormone-releasing Factor; AY 25650; AY-25650; AY25650; CL 118532; CL-118,532; CL-118532; CL118532; Detryptoreline
  Arms: Arm II (RT, ADT); Arm III (RT, ADT); Arm IV (RT, ADT, darolutamide)

SUMMARY:
This phase III trial uses the Decipher risk score to guide therapy selection. Decipher score is based on the activity of 22 genes in prostate tumor and may predict how likely it is for recurrent prostate cancer to spread (metastasize) to other parts of the body. Decipher score in this study is used for patient selection and the two variations of treatment to be studied: intensification for higher Decipher score or de-intensification for low Decipher score. Patients with higher Decipher risk score will be assigned to the part of the study that compares the use of 6 months of the usual treatment (hormone therapy and radiation treatment) to the use of darolutamide plus the usual treatment (intensification). The purpose of this section of the study is to determine whether the additional drug can reduce the chance of cancer coming back and spreading in patients with higher Decipher score. The addition of darolutamide to the usual treatment may better control the cancer and prevent it from spreading. Alternatively, patients with low Decipher risk score will be assigned to the part of the study that compares the use of radiation treatment alone (de-intensification) to the usual approach (6 months of hormone therapy plus radiation). The purpose of this part of the study is to determine if radiation treatment alone is as effective compared to the usual treatment without affecting the chance of tumor coming back in patients with low Decipher score prostate cancer. Radiation therapy uses high energy to kill tumor cells and reduce the tumor size. Hormone therapy drugs such as darolutamide suppress or block the production or action of male hormones that play role in prostate cancer development. Effect of radiation treatment alone in patients with low Decipher score prostate cancer could be the same as the usual approach in stabilizing prostate cancer and preventing it from spreading, while avoiding the side effects associated with hormonal therapy.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine whether men with National Comprehensive Cancer Network (NCCN) unfavorable intermediate risk (UIR) prostate cancer and lower Decipher genomic risk (Decipher score < 0.40) treated with radiation therapy (RT) alone instead of 6 months androgen deprivation therapy (ADT) + RT experience non-inferior rate of distant metastasis. (De-intensification study) II. To determine whether men with NCCN UIR prostate cancer who are in the higher genomic risk (Decipher score >= 0.40) will have a superior metastasis-free survival through treatment intensification with darolutamide added to the standard of RT plus 6 months ADT. (Intensification study)

SECONDARY OBJECTIVES:

I. To compare overall survival (OS) between the standard of care (RT plus 6 months of ADT) and either the de-intensification (RT alone) or intensification (RT plus 6 months of ADT plus darolutamide) interventions.

II. To compare time to prostate specific antigen (PSA) failure between the standard of care (RT plus 6 months of ADT) and either the de-intensification (RT alone) or intensification (RT plus 6 months of ADT plus darolutamide) interventions.

III. To compare metastasis free survival (MFS) based on conventional imaging between the standard of care (RT plus 6 months of ADT) and de-intensification intervention (RT alone).

IV. To compare MFS based on either conventional and/or molecular imaging between the standard of care (RT plus 6 months of ADT) and either the de-intensification (RT alone) or intensification (RT plus 6 months of ADT plus darolutamide) interventions.

V. To compare cumulative incidence of locoregional failure based upon conventional imaging and/ or biopsy between standard of care (RT plus 6 months of ADT) and either the de-intensification (RT alone) or intensification (RT plus 6 months ADT plus darolutamide) interventions.

VI. To compare cumulative incidence of distant metastasis based upon conventional imaging between standard of care (RT plus 6 months of ADT) and intensification intervention (RT plus 6 months ADT plus darolutamide).

VII. To compare cumulative incidence of distant metastasis based upon either conventional and/or molecular imaging between standard of care (RT plus 6 months of ADT) and either the de-intensification (RT alone) or intensification (RT plus 6 months of ADT plus darolutamide) interventions.

VIII. To compare prostate cancer-specific mortality between the standard of care (RT plus 6 months of ADT) and either the de-intensification (RT alone) or intensification (RT plus 6 months of ADT plus darolutamide) interventions.

IX. To compare sexual and hormonal related quality of life, as measured by the Expanded Prostate Cancer Index Composite-26 (EPIC), between the standard of care (RT plus 6 months of ADT) and either the de-intensification (RT alone) or intensification (RT plus 6 months of ADT plus darolutamide) interventions.

X. To compare fatigue, as measured by the Patient Reported Outcomes Measurement Information System (PROMIS)-Fatigue instrument, between the standard of care (RT plus 6 months of ADT) and either the de-intensification (RT alone) or intensification (RT plus 6 months of ADT plus darolutamide) interventions.

XI. To compare cognition, as measured by the Functional Assessment of Chronic Illness Therapy-Cognitive (FACT-Cog) perceived cognitive abilities subscale, between the standard of care (RT plus 6 months of ADT) and either the de-intensification (RT alone) or intensification (RT plus 6 months of ADT plus darolutamide) interventions.

EXPLORATORY OBJECTIVES:

I. To compare changes in cardio-metabolic markers, including body mass index, lipids, blood glucose, complete blood count (CBC), comprehensive metabolic panel (CMP), and hemoglobin (Hgb) A1c, between the standard of care (RT plus 6 months of ADT) and either the de-intensification (RT alone) or intensification (RT plus 6 months of ADT plus darolutamide) interventions.

II. To compare PSA failure-free survival with non-castrate testosterone and no additional therapies between the standard of care (RT plus 6 months of ADT) and either the de-intensification (RT alone) or intensification (RT plus 6 months of ADT plus darolutamide) interventions.

III. To compare cumulative incidence of locoregional failure based upon either conventional and/or molecular imaging between standard of care (RT plus 6 months of ADT) and either the de-intensification (RT alone) or intensification (RT plus 6 months of ADT plus darolutamide) interventions.

IV. To compare castrate-resistant prostate cancer (CRPC) between the standard of care (RT plus 6 months of ADT) and either the de-intensification (RT alone) or intensification (RT plus 6 months of ADT plus darolutamide) interventions.

V. To compare bowel and urinary function related quality of life, as measured by the Expanded Prostate Cancer Index Composite-26 (EPIC), between the standard of care (RT plus 6 months of ADT) and either the de-intensification (RT alone) or intensification (RT plus 6 months of ADT plus darolutamide) interventions.

VI. To compare time to testosterone recovery (defined as a T > 200ng/dL) between the standard of care (RT plus 6 months of ADT) and intensification (RT plus 6 months of ADT plus darolutamide) interventions.

VII. To compare health utilities, as measured by the European Quality of Life Five Dimension Five Level Scale (EQ-5D-5L), between the standard of care (RT plus 6 months of ADT) and either the de-intensification (RT alone) or intensification (RT plus 6 months of ADT plus darolutamide) interventions.

VIII. To develop and assess a machine learning/artificial intelligence algorithm for radiotherapy planning and/or quality assurance.

IX. To perform future translational correlative studies using biological data, Decipher results, and clinical outcomes.

OUTLINE:

DE-INTENSIFICATION STUDY: Patients with Decipher score < 0.40 are randomized to 1 of 2 arms.

ARM I: Patients undergo radiation therapy (RT) using a recognized regimen (2-3 days a week or 5 days a week for 2-11 weeks) in the absence of disease progression or unacceptable toxicity.

ARM II: Patients undergo RT as Arm I. Patients also receive androgen deprivation therapy (ADT) consisting of leuprolide, goserelin, buserelin, histrelin, triptorelin, degarelix, or relugolix at the discretion of the treating physician, for 6 months in the absence of disease progression or unacceptable toxicity. Patients may also receive bicalutamide or flutamide for 0, 30 or 180 days.

INTENSIFICATION STUDY: Patients with Decipher score >= 0.40 are randomized to 1 of 2 arms.

ARM III: Patients receive treatment as in Arm II.

ARM IV: Patients receive RT and ADT as in Arm II. Patients also receive darolutamide orally (PO) twice daily (BID). Treatment repeats every 90 days for up to 2 cycles in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 3, 6, 12, 24, 36, 48 and 60 months.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically (histologically or cytologically) proven diagnosis of adenocarcinoma of the prostate within 270 days prior to registration
* Unfavorable intermediate risk prostate cancer, defined as having ALL the following bulleted criteria:

  * Has at least one intermediate risk factor (IRF):

    * PSA 10-20 ng/mL
    * Clinical stage T2b-c (digital rectal examination [DRE] and/or imaging) by American Joint Committee on Cancer (AJCC) 8th edition
    * Gleason score 7 (Gleason 3+4 or 4+3 [ International Society of Urological Pathology (ISUP) Grade Group 2-3])
  * Has ONE or more of the following 'unfavorable' intermediate-risk designators:

    * > 1 immature reticulocyte fraction (IRF)
    * Gleason 4+3=7 (ISUP Grade Group 3)
    * >= 50% of biopsy cores positive

      * Biopsies may include 'sextant' sampling of right/left regions of the prostate, often labeled base, mid-gland and apex. All such 'sextant' biopsy cores should be counted. Men may also undergo 'targeted' sampling of prostate lesions (guided by MRI, ultrasound or other approaches). A targeted lesion that is biopsied more than once and demonstrates cancer (regardless of number of targeted cores involved) should count as a single additional positive core sampled and positive. In cases of uncertainty, count the biopsy sampling as sextant core(s)
  * Absence of high-risk features
* Appropriate stage for study entry based on the following diagnostic workup:

  * History/physical examination within 120 days prior to registration;
  * Negative bone imaging (M0) within 120 days prior to registration; Note: Tc-99m bone scan or sodium fluoride (NaF) positron emission tomography (PET) are allowed. Equivocal bone scan findings are allowed if plain films X-ray, computed tomography (CT) or magnetic resonance imaging (MRI) are negative for metastasis at the concerned site(s). While a negative fluciclovine, choline, or prostate specific membrane antigen (PSMA) PET may be counted as acceptable substitute for bone imaging, any suspicious findings must be confirmed and correlated with conventional imaging (Tc-99m bone scan, NaF PET, CT, X-ray, or MRI) to determine eligibility based on the latter modalities (e.g. M0 based on conventional imaging modalities)
  * Clinically negative lymph nodes (N0) as established by conventional imaging (pelvic +/- abdominal CT or MR), within 120 days prior to registration. Patients with lymph nodes equivocal or questionable by imaging are eligible if the nodes are =< 1.0 cm in short axis and/or if biopsy is negative.

Note: While a negative fluciclovine, choline, or prostate specific membrane antigen (PSMA) PET may be counted as acceptable substitute for pelvic imaging, any suspicious findings must be confirmed by conventional imaging (CT, MRI or biopsy). If the findings do not meet pathological criteria based on the latter modalities (e.g. node =< 10 mm in short axis, negative biopsy), the patient will still be eligible

* Age >= 18
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-2 within 120 days prior to registration
* Non-castrate testosterone level (> 50 ng/dL) within 120 days prior to registration
* Absolute neutrophil >= 1,000 cells/mm^3 (within 120 days prior to registration)
* Hemoglobin >= 8.0 g/dL, independent of transfusion and/or growth factors (within 120 days prior to registration)
* Platelet count >= 100,000 cells/mm^3 independent of transfusion and/or growth factors (within 120 days prior to registration)
* Creatinine clearance (CrCl) >= 30 mL/min estimated by Cockcroft-Gault equation (within 120 days prior to registration)

  * For African American patients specifically whose renal function is not considered adequate by the formula above, an alternative formula that takes race into account (Chronic Kidney Disease Epidemiology Collaboration CKD-EPI formula) should be used for calculating the related estimated glomerular filtration rate (GFR) with a correction factor for African American race creatinine clearance for trial eligibility, where GFR >= 30 mL/min/1.73m^2 will be considered adequate
* Total bilirubin: 1.5 =< institutional upper limit of normal (ULN) (within 120 days prior to registration) (Note: In subjects with Gilbert's syndrome, if total bilirubin is > 1.5 x ULN, measure direct and indirect bilirubin. If direct bilirubin is less than or equal to 1.5 x ULN, subject is eligible)
* Aspartate aminotransferase (AST)(serum glutamic-oxaloacetic transaminase [SGOT]) and alanine aminotransferase (ALT)(serum glutamate pyruvate transaminase [SGPT]): =< 2.5 x institutional ULN (within 120 days prior to registration)
* Human immunodeficiency virus (HIV)-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial; Note: HIV testing is not required for eligibility for this protocol
* For patients with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated.

  * Note: Known positive test for hepatitis B virus surface antigen (HBV sAg) indicating acute or chronic infection would make the patient ineligible unless the viral load becomes undetectable on suppressive therapy. Patients who are immune to hepatitis B (anti-Hepatitis B surface antibody positive) are eligible (e.g. patients immunized against hepatitis B)
* For patients with a history of hepatitis C virus (HCV) infection must have been treated and cured. For patients with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load

  * Note: Known positive test for hepatitis C virus ribonucleic acid (HCV RNA) indicating acute or chronic infection would make the patient ineligible unless the viral load becomes undetectable on suppressive therapy
* The patient or a legally authorized representative must provide study-specific informed consent prior to study entry and, for patients treated in the United States (U.S.), authorization permitting release of personal health information

Exclusion Criteria:

* Previous radical surgery (prostatectomy) or any form of curative-intent ablation whether focal or whole-gland (e.g., cryosurgery, high intensity focused ultrasound [HIFU], laser thermal ablation, etc.) for prostate cancer
* Definitive clinical or radiologic evidence of metastatic disease (M1)
* Prior invasive malignancy (except non-melanomatous skin cancer) unless disease free for a minimum of 3 years. History of or current diagnosis of hematologic malignancy is not allowed
* Prior radiotherapy to the prostate/pelvis region that would result in overlap of radiation therapy fields
* Previous bilateral orchiectomy
* Previous hormonal therapy, such as luteinizing hormone-releasing hormone (LHRH) agonists (e.g., leuprolide, goserelin, buserelin, triptorelin) or LHRH antagonist (e.g. degarelix), anti-androgens (e.g., flutamide, bicalutamide, cyproterone acetate). ADT started prior to study registration is not allowed
* Prior use of 5-alpha-reductase inhibitors is allowed, however, it must be stopped prior to enrollment on the study with at least a 30 day washout period before baseline study PSA measure and registration
* Active testosterone replacement therapy; any replacement therapy must be stopped at least 30 days prior to registration
* Severe, active co-morbidity defined as follows:

  * Current severe or unstable angina;
  * New York Heart Association Functional Classification III/IV (Note: Patients with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification)
  * History of any condition that in the opinion of the investigator, would preclude participation in this study
* Inability to swallow oral pills
* High risk features, which includes any of the following:

  * Gleason 8-10 [ISUP Grade Group 4-5]
  * PSA > 20
  * cT3-4 by digital exam OR gross extra-prostatic extension on imaging [indeterminate MRI evidence will not count and the patient will be eligible]

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2050 (Estimated)
Dates: Start 2021-12-06 (Actual); Primary Completion 2026-11-11 (Estimated); Study Completion 2026-11-11 (Estimated)

PRIMARY OUTCOMES:
Distant metastasis (DM) (De-intensification study) | From randomization to the detection of distant metastasis by conventional imaging, assessed up to 5 years
Metastasis-free survival (MFS) (Intensification study) | From randomization until the occurrence of distant metastasis by conventional imaging or death from any cause, assessed up to 5 years
  MFS will be estimated by the Kaplan-Meier (1958) method and compared between the two treatment arms using a stratified log-rank test (stratified by the randomization stratification factors) at one-sided alpha level of 0.025.

SECONDARY OUTCOMES:
Overall survival | From randomization to death from any cause, assessed up to 5 years
  Will be estimated by the Kaplan-Meier method and compared between treatments arms by stratified log-rank test. Cox regression models will also be fit, adjusted for the stratification factors, to estimate hazard ratios, together with 95% confidence intervals.
Time to prostate specific antigen (PSA) failure | Up to 5 years
  Defined as PSA > 2 ng/ml above the nadir post randomization. Will be analyzed using competing-risk methods (Gooley 1999) where, in each case, death prior to occurrence of the event in question will be a competing risk.
MFS (De-intensification study) | From randomization until the occurrence of distant metastasis by conventional imaging or death from any cause, assessed up to 5 years
  Will be estimated by the Kaplan-Meier method and compared between treatments arms by stratified log-rank test. Cox regression models will also be fit, adjusted for the stratification factors, to estimate hazard ratios, together with 95% confidence intervals.
MFS including positron emission tomography (PET) imaging | From randomization until the occurrence of distant metastasis by conventional and/or molecular imaging or death from any cause, assessed up to 5 years
  Will be estimated by the Kaplan-Meier method and compared between treatments arms by stratified log-rank test.
Locoregional failure (LRF) | From randomization until local or regional recurrence based upon conventional imaging or biopsy, assessed up to 5 years
  Will compare cumulative incidence between arms.
DM including PET imaging | From randomization to the detection of distant metastasis by conventional and/or molecular imaging, assessed up to 5 years
  Will be analyzed using competing-risk methods (Gooley 1999) where, in each case, death prior to occurrence of the event in question will be a competing risk.
Prostate cancer-specific mortality | From randomization until death from prostate cancer, assessed up to 5 years
  Will be analyzed using competing-risk methods (Gooley 1999) where, in each case death from causes other than prostate cancer as the competing risk.
Sexual and hormonal function related quality of life | Up to 5 years
  Measured by the Expanded Prostate Cancer Index Composite-26 (EPIC-26).
Fatigue | Up to 5 years
  Measured by the Patient Reported Outcomes Measurement Information System (PROMIS)-Fatigue instrument.
Cognition | Up to 5 years
  Measured by the Functional Assessment of Chronic illness Therapy-Cognitive (FACT-Cog).
DM (Intensification study) | From randomization to the detection of distant metastasis by conventional imaging, assessed up to 5 years
  Will be analyzed using competing-risk methods (Gooley 1999) where, in each case, death prior to occurrence of the event in question will be a competing risk.

OTHER OUTCOMES:
Castrate-resistant prostate cancer (CRPC) | Up to 5 years
  CRPC is defined as PSA increase > 25% and more than 2 ng/mL above nadir on study in conjunction with a serum testosterone (T) < 50 ng/mL, confirmed by repeat measurements at least 2 weeks apart. Will be analyzed using competing-risk methods (Gooley 1999) where, in each case, death prior to occurrence of the event in question will be a competing risk.
Bowel and urinary function related quality of life | Up to 5 years
  Measured EPIC-26. Mixed effect regression models will be fit to compare the changes over time in the domain scores. Covariates will include treatment, time, and treatment-by-time treatment interaction terms.
Cardio-metabolic markers | Up to 5 years
  Will include body mass index, lipids, blood glucose, complete blood count, comprehensive metabolic panel, and hemoglobin A1c. Mixed effect regression models will be fit to compare the changes over time in the cardio-metabolic markers between treatment groups. Covariates will include treatment, time, and treatment-by-time treatment interaction terms.
PSA failure-free survival with non-castrate testosterone and no additional therapies | Up to 5 years
Locoregional failure based upon either conventional or molecular imaging | Up to 5 years
Health utilities | Up to 5 years
  Measured by the European Quality of Life Five Dimension Five Level Scale (EQ-5D-5L). ). The bootstrap (Efron 1980) will be performed to obtain standard errors, test for significant differences, and generate 95% confidence intervals.
Time to testosterone recovery | From randomization until T > 200 ng/dL, assessed up to 5 years
  Will be analyzed using competing-risk methods (Gooley 1999) where, in each case, death prior to occurrence of the event in question will be a competing risk. Changes in quality of life measures will be correlated with changes in testosterone levels.

CONTACTS AND LOCATIONS:
Overall Officials: Neil B Desai, Principal Investigator — NRG Oncology
Locations (575):
- United States (566):
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - Banner MD Anderson Cancer Center, Gilbert, Arizona
  - Arizona Center for Cancer Care - Gilbert, Gilbert, Arizona
  - Arizona Center for Cancer Care-Peoria, Peoria, Arizona
  - Arizona Center for Cancer Care - Phoenix, Phoenix, Arizona
  - Arizona Center for Cancer Care - Scottsdale, Scottsdale, Arizona
  - Arizona Center for Cancer Care-Surprise, Surprise, Arizona
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Sutter Cancer Centers Radiation Oncology Services-Auburn, Auburn, California
  - AIS Cancer Center at San Joaquin Community Hospital, Bakersfield, California
  - Tower Cancer Research Foundation, Beverly Hills, California
  - Sutter Cancer Centers Radiation Oncology Services-Cameron Park, Cameron Park, California
  - City of Hope Corona, Corona, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Kaiser Permanente Dublin, Dublin, California
  - UC San Diego Health System - Encinitas, Encinitas, California
  - Kaiser Permanente-Fremont, Fremont, California
  - Washington Hospital, Fremont, California
  - Kaiser Permanente Fresno Orchard Plaza, Fresno, California
  - Kaiser Permanente-Fresno, Fresno, California
  - Marin General Hospital, Greenbrae, California
  - UCI Health - Chao Family Comprehensive Cancer Center and Ambulatory Care, Irvine, California
  - City of Hope at Irvine Lennar, Irvine, California
  - UC San Diego Moores Cancer Center, La Jolla, California
  - City of Hope Antelope Valley, Lancaster, California
  - Los Angeles General Medical Center, Los Angeles, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - Fremont - Rideout Cancer Center, Marysville, California
  - Memorial Medical Center, Modesto, California
  - Kaiser Permanente-Modesto, Modesto, California
  - Providence Queen of The Valley, Napa, California
  - Kaiser Permanente-Oakland, Oakland, California
  - Saint Joseph Hospital - Orange, Orange, California
  - UC Irvine Health/Chao Family Comprehensive Cancer Center, Orange, California
  - Palo Alto Medical Foundation Health Care, Palo Alto, California
  - Kaiser Permanente-Roseville, Roseville, California
  - Sutter Cancer Centers Radiation Oncology Services-Roseville, Roseville, California
  - Kaiser Permanente Downtown Commons, Sacramento, California
  - Sutter Medical Center Sacramento, Sacramento, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Kaiser Permanente-South Sacramento, Sacramento, California
  - California Protons Cancer Therapy Center, San Diego, California
  - Sharp Memorial Hospital, San Diego, California
  - Kaiser Permanente-San Francisco, San Francisco, California
  - UCSF Medical Center-Mission Bay, San Francisco, California
  - Kaiser Permanente-Santa Teresa-San Jose, San Jose, California
  - Kaiser Permanente San Leandro, San Leandro, California
  - Ridley-Tree Cancer Center, Santa Barbara, California
  - Kaiser Permanente Medical Center - Santa Clara, Santa Clara, California
  - Kaiser Permanente-Santa Rosa, Santa Rosa, California
  - City of Hope South Pasadena, South Pasadena, California
  - Kaiser Permanente-South San Francisco, South San Francisco, California
  - Palo Alto Medical Foundation-Sunnyvale, Sunnyvale, California
  - Cedars-Sinai Cancer - Tarzana, Tarzana, California
  - City of Hope South Bay, Torrance, California
  - Torrance Memorial Physician Network - Cancer Care, Torrance, California
  - Torrance Memorial Medical Center, Torrance, California
  - Gene Upshaw Memorial Tahoe Forest Cancer Center, Truckee, California
  - City of Hope Upland, Upland, California
  - Kaiser Permanente-Vallejo, Vallejo, California
  - Sutter Solano Medical Center/Cancer Center, Vallejo, California
  - Kaiser Permanente-Walnut Creek, Walnut Creek, California
  - BASS Medical Group - Lennon, Walnut Creek, California
  - UCHealth University of Colorado Hospital, Aurora, Colorado
  - Rocky Mountain Cancer Centers-Boulder, Boulder, Colorado
  - UCHealth Memorial Hospital Central, Colorado Springs, Colorado
  - Memorial Hospital North, Colorado Springs, Colorado
  - Shaw Cancer Center, Edwards, Colorado
  - Poudre Valley Hospital, Fort Collins, Colorado
  - Cancer Care and Hematology-Fort Collins, Fort Collins, Colorado
  - Banner North Colorado Medical Center, Greeley, Colorado
  - UCHealth Greeley Hospital, Greeley, Colorado
  - UCHealth Highlands Ranch Hospital, Highlands Ranch, Colorado
  - Medical Center of the Rockies, Loveland, Colorado
  - Banner North Colorado Medical Center - Loveland Campus, Loveland, Colorado
  - Hartford HealthCare - Saint Vincent's Medical Center, Bridgeport, Connecticut
  - Danbury Hospital, Danbury, Connecticut
  - Smilow Cancer Hospital Care Center at Greenwich, Greenwich, Connecticut
  - Smilow Cancer Hospital Care Center - Guilford, Guilford, Connecticut
  - Hartford Hospital, Hartford, Connecticut
  - Midstate Medical Center, Meriden, Connecticut
  - The Hospital of Central Connecticut, New Britain, Connecticut
  - Yale University, New Haven, Connecticut
  - Norwalk Hospital, Norwalk, Connecticut
  - Smilow Cancer Hospital Care Center-Trumbull, Trumbull, Connecticut
  - Smilow Cancer Hospital Care Center - Waterford, Waterford, Connecticut
  - Beebe South Coastal Health Campus, Millville, Delaware
  - Helen F Graham Cancer Center, Newark, Delaware
  - Medical Oncology Hematology Consultants PA, Newark, Delaware
  - Beebe Health Campus, Rehoboth Beach, Delaware
  - George Washington University Medical Center, Washington D.C., District of Columbia
  - Bay Pines VA Healthcare System, Bay Pines, Florida
  - Boca Raton Regional Hospital, Boca Raton, Florida
  - UF Health Cancer Institute - Gainesville, Gainesville, Florida
  - Jupiter Medical Center, Jupiter, Florida
  - GenesisCare USA - Plantation, Plantation, Florida
  - Cleveland Clinic-Weston, Weston, Florida
  - Grady Health System, Atlanta, Georgia
  - Emory Proton Therapy Center, Atlanta, Georgia
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Piedmont Hospital, Atlanta, Georgia
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Emory Saint Joseph's Hospital, Atlanta, Georgia
  - Emory Decatur Hospital, Decatur, Georgia
  - Piedmont Fayette Hospital, Fayetteville, Georgia
  - Northeast Georgia Medical Center-Gainesville, Gainesville, Georgia
  - Emory Johns Creek Hospital, Johns Creek, Georgia
  - Lewis Cancer and Research Pavilion at Saint Joseph's/Candler, Savannah, Georgia
  - Hawaii Cancer Care Inc - Waterfront Plaza, Honolulu, Hawaii
  - Queen's Cancer Cenrer - POB I, Honolulu, Hawaii
  - Queen's Medical Center, Honolulu, Hawaii
  - Straub Clinic and Hospital, Honolulu, Hawaii
  - Queen's Cancer Center - Kuakini, Honolulu, Hawaii
  - The Cancer Center of Hawaii-Liliha, Honolulu, Hawaii
  - Hawaii Cancer Care - Westridge, ‘Aiea, Hawaii
  - Pali Momi Medical Center, ‘Aiea, Hawaii
  - The Queen's Medical Center - West Oahu, ‘Ewa Beach, Hawaii
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - Saint Luke's Cancer Institute - Fruitland, Fruitland, Idaho
  - Saint Luke's Cancer Institute - Meridian, Meridian, Idaho
  - Saint Luke's Cancer Institute - Nampa, Nampa, Idaho
  - Saint Luke's Cancer Institute - Twin Falls, Twin Falls, Idaho
  - Alton Memorial Hospital, Alton, Illinois
  - Rush-Copley Medical Center, Aurora, Illinois
  - Advocate Good Shepherd Hospital, Barrington, Illinois
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Northwestern University, Chicago, Illinois
  - Rush MD Anderson Cancer Center, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - Advocate Illinois Masonic Medical Center, Chicago, Illinois
  - AMG Crystal Lake - Oncology, Crystal Lake, Illinois
  - Carle at The Riverfront, Danville, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Northwestern Medicine Cancer Center Kishwaukee, DeKalb, Illinois
  - Advocate Good Samaritan Hospital, Downers Grove, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Advocate Sherman Hospital, Elgin, Illinois
  - Elmhurst Memorial Hospital, Elmhurst, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Northwestern Medicine Cancer Center Delnor, Geneva, Illinois
  - Northwestern Medicine Glenview Outpatient Center, Glenview, Illinois
  - Northwestern Medicine Grayslake Outpatient Center, Grayslake, Illinois
  - Advocate South Suburban Hospital, Hazel Crest, Illinois
  - Edward Hines Jr VA Hospital, Hines, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - Northwestern Medicine Lake Forest Hospital, Lake Forest, Illinois
  - AMG Libertyville - Oncology, Libertyville, Illinois
  - Condell Memorial Hospital, Libertyville, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Edward Hospital/Cancer Center, Naperville, Illinois
  - HSHS Saint Elizabeth's Hospital, O'Fallon, Illinois
  - Northwestern Medicine Oak Brook, Oak Brook, Illinois
  - Advocate Christ Medical Center, Oak Lawn, Illinois
  - Northwestern Medicine Orland Park, Orland Park, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Advocate High Tech Medical Park, Palos Heights, Illinois
  - Advocate Lutheran General Hospital, Park Ridge, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - UW Health Carbone Cancer Center Rockford, Rockford, Illinois
  - Memorial Hospital East, Shiloh, Illinois
  - Springfield Memorial Hospital, Springfield, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - Northwestern Medicine Cancer Center Warrenville, Warrenville, Illinois
  - Illinois CancerCare - Washington, Washington, Illinois
  - Saint Luke's Hospital, Cedar Rapids, Iowa
  - Mercy Hospital, Cedar Rapids, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - University of Kansas Cancer Center, Kansas City, Kansas
  - The University of Kansas Cancer Center - Olathe, Olathe, Kansas
  - University of Kansas Cancer Center-Overland Park, Overland Park, Kansas
  - University of Kansas Hospital-Indian Creek Campus, Overland Park, Kansas
  - Salina Regional Health Center, Salina, Kansas
  - Cotton O'Neil Cancer Center / Stormont Vail Health, Topeka, Kansas
  - University of Kansas Health System Saint Francis Campus, Topeka, Kansas
  - University of Kansas Hospital-Westwood Cancer Center, Westwood, Kansas
  - Ascension Via Christi Hospitals Wichita, Wichita, Kansas
  - Saint Joseph Radiation Oncology Resource Center, Lexington, Kentucky
  - Mary Bird Perkins Cancer Center - Metairie, Metairie, Louisiana
  - East Jefferson General Hospital, Metairie, Louisiana
  - LSU Healthcare Network / Metairie Multi-Specialty Clinic, Metairie, Louisiana
  - MaineHealth Maine Medical Center - Portland, Portland, Maine
  - Penobscot Bay Medical Center, Rockport, Maine
  - MaineHealth Maine Medical Center- Scarborough, Scarborough, Maine
  - MaineHealth Cancer Care and IV Therapy - South Portland, South Portland, Maine
  - Luminis Health Anne Arundel Medical Center, Annapolis, Maryland
  - Maryland Proton Treatment Center, Baltimore, Maryland
  - University of Maryland/Greenebaum Cancer Center, Baltimore, Maryland
  - UM Upper Chesapeake Medical Center, Bel Air, Maryland
  - Central Maryland Radiation Oncology in Howard County, Columbia, Maryland
  - University of Maryland Shore Medical Center at Easton, Easton, Maryland
  - UM Baltimore Washington Medical Center/Tate Cancer Center, Glen Burnie, Maryland
  - UM Capital Region Medical Center, Largo, Maryland
  - TidalHealth Richard A Henson Cancer Institute, Ocean Pines, Maryland
  - TidalHealth Peninsula Regional, Salisbury, Maryland
  - Beverly Hospital, Beverly, Massachusetts
  - Lahey Hospital and Medical Center, Burlington, Massachusetts
  - Addison Gilbert Hospital, Gloucester, Massachusetts
  - Lahey Medical Center-Peabody, Peabody, Massachusetts
  - Beth Israel Deaconess Medical Center/Winchester Center for Cancer Care, Winchester, Massachusetts
  - Veteran's Administration Medical Center - Ann Arbor, Ann Arbor, Michigan
  - Trinity Health Saint Joseph Mercy Hospital Ann Arbor, Ann Arbor, Michigan
  - University of Michigan Rogel Cancer Center, Ann Arbor, Michigan
  - McLaren Cancer Institute-Bay City, Bay City, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Brighton, Brighton, Michigan
  - Trinity Health Medical Center - Brighton, Brighton, Michigan
  - Henry Ford Cancer Institute-Downriver, Brownstown, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Canton, Canton, Michigan
  - Trinity Health Medical Center - Canton, Canton, Michigan
  - Chelsea Hospital, Chelsea, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Chelsea Hospital, Chelsea, Michigan
  - McLaren Cancer Institute-Clarkston, Clarkston, Michigan
  - Michigan Healthcare Professionals Clarkston, Clarkston, Michigan
  - Henry Ford Macomb Hospital-Clinton Township, Clinton Township, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Michigan Healthcare Professionals Farmington, Farmington Hills, Michigan
  - Weisberg Cancer Treatment Center, Farmington Hills, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - McLaren Cancer Institute-Flint, Flint, Michigan
  - Trinity Health Grand Rapids Hospital, Grand Rapids, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Karmanos Cancer Institute at McLaren Greater Lansing, Lansing, Michigan
  - University of Michigan Health - Sparrow Lansing, Lansing, Michigan
  - McLaren Cancer Institute-Lapeer Region, Lapeer, Michigan
  - Trinity Health Saint Mary Mercy Livonia Hospital, Livonia, Michigan
  - Michigan Healthcare Professionals Macomb, Macomb, Michigan
  - Michigan Healthcare Professionals Madison Heights, Madison Heights, Michigan
  - McLaren Cancer Institute-Macomb, Mount Clemens, Michigan
  - McLaren Cancer Institute-Central Michigan, Mount Pleasant, Michigan
  - Corewell Health Lakeland Hospitals - Niles Hospital, Niles, Michigan
  - Henry Ford Medical Center-Columbus, Novi, Michigan
  - McLaren Cancer Institute-Northern Michigan, Petoskey, Michigan
  - Trinity Health Saint Joseph Mercy Oakland Hospital, Pontiac, Michigan
  - McLaren-Port Huron, Port Huron, Michigan
  - Corewell Health William Beaumont University Hospital, Royal Oak, Michigan
  - MyMichigan Medical Center Saginaw, Saginaw, Michigan
  - Corewell Health Lakeland Hospitals - Marie Yeager Cancer Center, Saint Joseph, Michigan
  - Corewell Health Lakeland Hospitals - Saint Joseph Hospital, Saint Joseph, Michigan
  - MyMichigan Medical Center Tawas, Tawas City, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - Corewell Health Beaumont Troy Hospital, Troy, Michigan
  - Michigan Healthcare Professionals Troy, Troy, Michigan
  - Henry Ford West Bloomfield Hospital, West Bloomfield, Michigan
  - University of Michigan Health - West, Wyoming, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology Ann Arbor Campus, Ypsilanti, Michigan
  - Mercy Hospital, Coon Rapids, Minnesota
  - Miller-Dwan Hospital, Duluth, Minnesota
  - Saint Luke's Hospital of Duluth, Duluth, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Siteman Cancer Center at Saint Peters Hospital, City of Saint Peters, Missouri
  - MU Health - University Hospital/Ellis Fischel Cancer Center, Columbia, Missouri
  - Siteman Cancer Center at West County Hospital, Creve Coeur, Missouri
  - Parkland Health Center - Farmington, Farmington, Missouri
  - University of Kansas Cancer Center - Briarcliff, Kansas City, Missouri
  - University of Kansas Cancer Center - North, Kansas City, Missouri
  - University of Kansas Cancer Center - Lee's Summit, Lee's Summit, Missouri
  - University of Kansas Cancer Center at North Kansas City Hospital, North Kansas City, Missouri
  - Phelps Health Delbert Day Cancer Institute, Rolla, Missouri
  - Sainte Genevieve County Memorial Hospital, Sainte Genevieve, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - SSM Health Saint Louis University Hospital, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Siteman Cancer Center-South County, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Siteman Cancer Center at Christian Hospital, St Louis, Missouri
  - Missouri Baptist Sullivan Hospital, Sullivan, Missouri
  - BJC Outpatient Center at Sunset Hills, Sunset Hills, Missouri
  - Billings Clinic Cancer Center, Billings, Montana
  - Saint James Community Hospital and Cancer Treatment Center, Butte, Montana
  - Benefis Sletten Cancer Institute, Great Falls, Montana
  - Nebraska Medicine-Bellevue, Bellevue, Nebraska
  - Nebraska Medicine-Village Pointe, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - New Hampshire Oncology Hematology PA-Concord, Concord, New Hampshire
  - Dartmouth Hitchcock Medical Center/Dartmouth Cancer Center, Lebanon, New Hampshire
  - Solinsky Center for Cancer Care, Manchester, New Hampshire
  - Memorial Sloan Kettering Basking Ridge, Basking Ridge, New Jersey
  - Clara Maass Medical Center, Belleville, New Jersey
  - Cooper Hospital University Medical Center, Camden, New Jersey
  - AtlantiCare Surgery Center, Egg Harbor, New Jersey
  - Trinitas Hospital and Comprehensive Cancer Center - Williamson Street Campus, Elizabeth, New Jersey
  - Englewood Hospital and Medical Center, Englewood, New Jersey
  - The Cancer Institute of New Jersey Hamilton, Hamilton, New Jersey
  - Jersey City Medical Center, Jersey City, New Jersey
  - Saint Barnabas Medical Center, Livingston, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Bergen, Montvale, New Jersey
  - Cooper CyberKnife Center, Mount Laurel, New Jersey
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Rutgers New Jersey Medical School, Newark, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - The Valley Hospital - Luckow Pavilion, Paramus, New Jersey
  - Sidney Kimmel Cancer Center Washington Township, Sewell, New Jersey
  - Robert Wood Johnson University Hospital Somerset, Somerville, New Jersey
  - Community Medical Center, Toms River, New Jersey
  - MD Anderson Cancer Center at Cooper-Voorhees, Voorhees Township, New Jersey
  - Lovelace Medical Center-Saint Joseph Square, Albuquerque, New Mexico
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Lovelace Radiation Oncology, Albuquerque, New Mexico
  - Presbyterian Kaseman Hospital, Albuquerque, New Mexico
  - Presbyterian Rust Medical Center/Jorgensen Cancer Center, Rio Rancho, New Mexico
  - Northwell Health Imbert Cancer Center, Bay Shore, New York
  - New York-Presbyterian/Brooklyn Methodist Hospital, Brooklyn, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - Memorial Sloan Kettering Commack, Commack, New York
  - Mary Imogene Bassett Hospital, Cooperstown, New York
  - Noyes Memorial Hospital/Myers Cancer Center, Dansville, New York
  - Arnot Ogden Medical Center/Falck Cancer Center, Elmira, New York
  - The New York Hospital Medical Center of Queens, Flushing, New York
  - Northwell Health Physicians Partners Radiation Medicine at Queens, Forest Hills, New York
  - Glens Falls Hospital, Glens Falls, New York
  - Northwell Health Cancer Institute at Huntington, Greenlawn, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Northwell Health/Center for Advanced Medicine, Lake Success, New York
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - Manhattan Eye Ear and Throat Hospital, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Lenox Hill Hospital, New York, New York
  - Queens Cancer Center, Rego Park, New York
  - Highland Hospital, Rochester, New York
  - University of Rochester, Rochester, New York
  - Phelps Memorial Hospital Center, Sleepy Hollow, New York
  - Staten Island University Hospital, Staten Island, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - Montefiore Medical Center-Einstein Campus, The Bronx, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - Memorial Sloan Kettering Nassau, Uniondale, New York
  - Westchester Medical Center, Valhalla, New York
  - Wilmot Cancer Institute at Webster, Webster, New York
  - Mission Hospital, Asheville, North Carolina
  - Duke Cancer Center Cary, Cary, North Carolina
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Durham VA Medical Center, Durham, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - UNC Health Cancer Care Raleigh, Raleigh, North Carolina
  - Duke Cancer Center Raleigh, Raleigh, North Carolina
  - UNC Health Cancer Care Wakefield, Raleigh, North Carolina
  - Novant Cancer Institute Radiation Oncology - Supply, Supply, North Carolina
  - Novant Health Cancer Institute Radiation Oncology - Wilmington, Wilmington, North Carolina
  - Novant Health New Hanover Regional Medical Center, Wilmington, North Carolina
  - Sanford Bismarck Medical Center, Bismarck, North Dakota
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Sanford Roger Maris Cancer Center, Fargo, North Dakota
  - Altru Cancer Center, Grand Forks, North Dakota
  - Summa Health System - Akron Campus, Akron, Ohio
  - Cleveland Clinic Akron General, Akron, Ohio
  - UH Seidman Cancer Center at UH Avon Health Center, Avon, Ohio
  - Summa Health System - Barberton Campus, Barberton, Ohio
  - UHHS-Chagrin Highlands Medical Center, Beachwood, Ohio
  - Aultman Health Foundation, Canton, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - University of Cincinnati Cancer Center-UC Medical Center, Cincinnati, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio
  - Cleveland Clinic Cancer Center/Fairview Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Grant Medical Center, Columbus, Ohio
  - Doctors Hospital, Columbus, Ohio
  - Delaware Health Center-Grady Cancer Center, Delaware, Ohio
  - Dublin Methodist Hospital, Dublin, Ohio
  - OhioHealth Mansfield Hospital, Mansfield, Ohio
  - Cleveland Clinic Cancer Center Mansfield, Mansfield, Ohio
  - OhioHealth Marion General Hospital, Marion, Ohio
  - Hillcrest Hospital Cancer Center, Mayfield Heights, Ohio
  - Summa Health Medina Medical Center, Medina, Ohio
  - UH Seidman Cancer Center at Lake Health Mentor Campus, Mentor, Ohio
  - UH Seidman Cancer Center at Southwest General Hospital, Middleburg Heights, Ohio
  - University Hospitals Parma Medical Center, Parma, Ohio
  - University Hospitals Portage Medical Center, Ravenna, Ohio
  - North Coast Cancer Care, Sandusky, Ohio
  - UH Seidman Cancer Center at Firelands Regional Medical Center, Sandusky, Ohio
  - Cleveland Clinic Cancer Center Strongsville, Strongsville, Ohio
  - ProMedica Flower Hospital, Sylvania, Ohio
  - South Pointe Hospital, Warrensville Heights, Ohio
  - University of Cincinnati Cancer Center-West Chester, West Chester, Ohio
  - Cleveland Clinic Wooster Family Health and Surgery Center, Wooster, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Saint Charles Health System, Bend, Oregon
  - Legacy Mount Hood Medical Center, Gresham, Oregon
  - Legacy Good Samaritan Hospital and Medical Center, Portland, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - Legacy Meridian Park Hospital, Tualatin, Oregon
  - Saint Luke's Cancer Center - Allentown, Allentown, Pennsylvania
  - UPMC Altoona, Altoona, Pennsylvania
  - UPMC-Heritage Valley Health System Beaver, Beaver, Pennsylvania
  - Saint Luke's University Hospital-Bethlehem Campus, Bethlehem, Pennsylvania
  - Crozer-Keystone Regional Cancer Center at Broomall, Broomall, Pennsylvania
  - Carlisle Regional Cancer Center, Carlisle, Pennsylvania
  - Christiana Care Health System-Concord Health Center, Chadds Ford, Pennsylvania
  - Chambersburg Hospital, Chambersburg, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Delaware County Memorial Hospital, Drexel Hill, Pennsylvania
  - Northeast Radiation Oncology Center, Dunmore, Pennsylvania
  - Saint Luke's Hospital-Anderson Campus, Easton, Pennsylvania
  - Ephrata Cancer Center, Ephrata, Pennsylvania
  - UPMC Hillman Cancer Center Erie, Erie, Pennsylvania
  - Saint Vincent Hospital, Erie, Pennsylvania
  - UPMC Cancer Center at UPMC Horizon, Farrell, Pennsylvania
  - Adams Cancer Center, Gettysburg, Pennsylvania
  - Crozer Regional Cancer Center at Brinton Lake, Glen Mills, Pennsylvania
  - UPMC Cancer Centers - Arnold Palmer Pavilion, Greensburg, Pennsylvania
  - UPMC Pinnacle Cancer Center/Community Osteopathic Campus, Harrisburg, Pennsylvania
  - Penn State Milton S Hershey Medical Center, Hershey, Pennsylvania
  - IRMC Cancer Center, Indiana, Pennsylvania
  - Jefferson Hospital, Jefferson Hills, Pennsylvania
  - UPMC-Johnstown/John P. Murtha Regional Cancer Center, Johnstown, Pennsylvania
  - Sechler Family Cancer Center, Lebanon, Pennsylvania
  - Geisinger Medical Oncology-Lewisburg, Lewisburg, Pennsylvania
  - Yolanda G Barco Oncology Institute, Meadville, Pennsylvania
  - UPMC Hillman Cancer Center at Rocco And Nancy Ortenzio Cancer Pavilion, Mechanicsburg, Pennsylvania
  - Forbes Hospital, Monroeville, Pennsylvania
  - UPMC Cancer Center - Monroeville, Monroeville, Pennsylvania
  - UPMC Hillman Cancer Center - Monroeville, Monroeville, Pennsylvania
  - UPMC Hillman Cancer Center in Coraopolis, Moon Township, Pennsylvania
  - Allegheny Valley Hospital, Natrona Heights, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Jefferson Torresdale Hospital, Philadelphia, Pennsylvania
  - Einstein Medical Center Philadelphia, Philadelphia, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - UPMC-Saint Margaret, Pittsburgh, Pennsylvania
  - West Penn Hospital, Pittsburgh, Pennsylvania
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - UPMC-Shadyside Hospital, Pittsburgh, Pennsylvania
  - UPMC-Passavant Hospital, Pittsburgh, Pennsylvania
  - UPMC-Saint Clair Hospital Cancer Center, Pittsburgh, Pennsylvania
  - Geisinger Cancer Services-Pottsville, Pottsville, Pennsylvania
  - Saint Luke's Hospital - Upper Bucks Campus, Quakertown, Pennsylvania
  - Saint Luke's Hospital-Quakertown Campus, Quakertown, Pennsylvania
  - UPMC Cancer Center at UPMC Northwest, Seneca, Pennsylvania
  - Saint Luke's Hospital - Monroe Campus, Stroudsburg, Pennsylvania
  - UPMC Cancer Center-Washington, Washington, Pennsylvania
  - UPMC Washington Hospital Radiation Oncology, Washington, Pennsylvania
  - Chester County Hospital, West Chester, Pennsylvania
  - Reading Hospital, West Reading, Pennsylvania
  - Wexford Health and Wellness Pavilion, Wexford, Pennsylvania
  - Geisinger Wyoming Valley/Henry Cancer Center, Wilkes-Barre, Pennsylvania
  - Divine Providence Hospital, Williamsport, Pennsylvania
  - Asplundh Cancer Pavilion, Willow Grove, Pennsylvania
  - WellSpan Health-York Cancer Center, York, Pennsylvania
  - UPMC Memorial, York, Pennsylvania
  - Saint Joseph's/Candler - Bluffton Campus, Bluffton, South Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - MUSC Health Florence Medical Center, Florence, South Carolina
  - Saint Francis Hospital, Greenville, South Carolina
  - Saint Francis Cancer Center, Greenville, South Carolina
  - Self Regional Healthcare, Greenwood, South Carolina
  - Gibbs Cancer Center-Pelham, Greer, South Carolina
  - The Radiation Oncology Center-Hilton Head/Bluffton, Hilton Head Island, South Carolina
  - Carolina Regional Cancer Center, Myrtle Beach, South Carolina
  - Beaufort Memorial/New River Cancer Center, Okatie, South Carolina
  - Spartanburg Medical Center, Spartanburg, South Carolina
  - Sanford Cancer Center Oncology Clinic, Sioux Falls, South Dakota
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - The Children's Hospital at TriStar Centennial, Nashville, Tennessee
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - MD Anderson in The Woodlands, Conroe, Texas
  - Parkland Memorial Hospital, Dallas, Texas
  - UT Southwestern Simmons Cancer Center - RedBird, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - Brooke Army Medical Center, Fort Sam Houston, Texas
  - UT Southwestern/Simmons Cancer Center-Fort Worth, Fort Worth, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - MD Anderson West Houston, Houston, Texas
  - MD Anderson League City, League City, Texas
  - UT Southwestern Clinical Center at Richardson/Plano, Richardson, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - MD Anderson in Sugar Land, Sugar Land, Texas
  - American Fork Hospital / Huntsman Intermountain Cancer Center, American Fork, Utah
  - Sandra L Maxwell Cancer Center, Cedar City, Utah
  - Farmington Health Center, Farmington, Utah
  - Logan Regional Hospital, Logan, Utah
  - Intermountain Medical Center, Murray, Utah
  - McKay-Dee Hospital Center, Ogden, Utah
  - Utah Valley Regional Medical Center, Provo, Utah
  - Riverton Hospital, Riverton, Utah
  - University of Utah Sugarhouse Health Center, Salt Lake City, Utah
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - LDS Hospital, Salt Lake City, Utah
  - Saint George Regional Medical Center, St. George, Utah
  - Central Vermont Medical Center/National Life Cancer Treatment, Berlin Corners, Vermont
  - University of Vermont Medical Center, Burlington, Vermont
  - Dartmouth Cancer Center - North, Saint Johnsbury, Vermont
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - Inova Schar Cancer Institute, Fairfax, Virginia
  - Inova Fair Oaks Hospital, Fairfax, Virginia
  - Bon Secours Saint Francis Medical Center, Midlothian, Virginia
  - Bon Secours Cancer Institute at Reynolds Crossing, Richmond, Virginia
  - VCU Massey Comprehensive Cancer Center, Richmond, Virginia
  - Virginia Mason Medical Center, Seattle, Washington
  - Legacy Cancer Institute Medical Oncology and Day Treatment, Vancouver, Washington
  - Legacy Salmon Creek Hospital, Vancouver, Washington
  - Providence Saint Mary Regional Cancer Center, Walla Walla, Washington
  - Langlade Hospital and Cancer Center, Antigo, Wisconsin
  - ThedaCare Regional Cancer Center, Appleton, Wisconsin
  - Ascension Saint Elizabeth Hospital, Appleton, Wisconsin
  - Northwest Wisconsin Cancer Center, Ashland, Wisconsin
  - Ascension Southeast Wisconsin Hospital - Elmbrook Campus, Brookfield, Wisconsin
  - Aurora Cancer Care-Southern Lakes VLCC, Burlington, Wisconsin
  - Ascension Calumet Hospital, Chilton, Wisconsin
  - Marshfield Medical Center-EC Cancer Center, Eau Claire, Wisconsin
  - Ascension Saint Francis - Reiman Cancer Center, Franklin, Wisconsin
  - Aurora Health Care Germantown Health Center, Germantown, Wisconsin
  - Aurora Cancer Care-Grafton, Grafton, Wisconsin
  - Bellin Memorial Hospital, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center at Saint Mary's, Green Bay, Wisconsin
  - Aurora BayCare Medical Center, Green Bay, Wisconsin
  - University of Wisconsin Carbone Cancer Center - Johnson Creek, Johnson Creek, Wisconsin
  - Aurora Cancer Care-Kenosha South, Kenosha, Wisconsin
  - University of Wisconsin Carbone Cancer Center - Eastpark Medical Center, Madison, Wisconsin
  - University of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin
  - Aurora Bay Area Medical Group-Marinette, Marinette, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Froedtert Menomonee Falls Hospital, Menomonee Falls, Wisconsin
  - Ascension Columbia Saint Mary's Hospital Ozaukee, Mequon, Wisconsin
  - Aurora Cancer Care-Milwaukee, Milwaukee, Wisconsin
  - Ascension Columbia Saint Mary's Hospital - Milwaukee, Milwaukee, Wisconsin
  - Aurora Saint Luke's Medical Center, Milwaukee, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Aurora Sinai Medical Center, Milwaukee, Wisconsin
  - Zablocki Veterans Administration Medical Center, Milwaukee, Wisconsin
  - Marshfield Medical Center - Minocqua, Minocqua, Wisconsin
  - ProHealth D N Greenwald Center, Mukwonago, Wisconsin
  - Drexel Town Square Health Center, Oak Creek, Wisconsin
  - ProHealth Oconomowoc Memorial Hospital, Oconomowoc, Wisconsin
  - Ascension Mercy Hospital, Oshkosh, Wisconsin
  - Vince Lombardi Cancer Clinic - Oshkosh, Oshkosh, Wisconsin
  - Ascension All Saints Hospital, Racine, Wisconsin
  - Aurora Cancer Care-Racine, Racine, Wisconsin
  - Aspirus Cancer Care - James Beck Cancer Center, Rhinelander, Wisconsin
  - Marshfield Medical Center-Rice Lake, Rice Lake, Wisconsin
  - Saint Vincent Hospital Cancer Center at Sheboygan, Sheboygan, Wisconsin
  - Vince Lombardi Cancer Clinic-Sheboygan, Sheboygan, Wisconsin
  - Aspirus Cancer Care - Stevens Point, Stevens Point, Wisconsin
  - Marshfield Medical Center-River Region at Stevens Point, Stevens Point, Wisconsin
  - Saint Vincent Hospital Cancer Center at Sturgeon Bay, Sturgeon Bay, Wisconsin
  - Aurora Medical Center in Summit, Summit, Wisconsin
  - Vince Lombardi Cancer Clinic-Two Rivers, Two Rivers, Wisconsin
  - UW Cancer Center at ProHealth Care, Waukesha, Wisconsin
  - Aspirus Regional Cancer Center, Wausau, Wisconsin
  - Ascension Medical Group Southeast Wisconsin - Mayfair Road, Wauwatosa, Wisconsin
  - Aurora Cancer Care-Milwaukee West, Wauwatosa, Wisconsin
  - Aurora West Allis Medical Center, West Allis, Wisconsin
  - Froedtert West Bend Hospital/Kraemer Cancer Center, West Bend, Wisconsin
  - Marshfield Medical Center - Weston, Weston, Wisconsin
  - Aspirus Cancer Care - Wisconsin Rapids, Wisconsin Rapids, Wisconsin
- Canada (9):
  - Arthur J E Child Comprehensive Cancer Centre, Calgary, Alberta
  - Atlantic Health Sciences Corporation-Saint John Regional Hospital, Saint John, New Brunswick
  - Juravinski Cancer Centre at Hamilton Health Sciences, Hamilton, Ontario
  - University Health Network-Princess Margaret Hospital, Toronto, Ontario
  - The Research Institute of the McGill University Health Centre (MUHC), Montreal, Quebec
  - CHU de Quebec-L'Hotel-Dieu de Quebec (HDQ), Québec, Quebec
  - Centre Hospitalier Universitaire de Sherbrooke-Fleurimont, Sherbrooke, Quebec
  - Allan Blair Cancer Centre, Regina, Saskatchewan
  - Saskatoon Cancer Centre, Saskatoon, Saskatchewan